CLINICAL TRIAL: NCT00733512
Title: Surgeon Experience ReSTOR Aspheric +4 Intraocular Lens (IOL)
Brief Title: Surgeon Experience ReSTOR A +4 Intraocular Lens (IOL)
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: M07-019
Record Dates: First submitted 2008-08-08; First posted 2008-08-13 (Estimated); Results first posted 2010-04-15 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2010-04

CONDITIONS: Cataract
Keywords: ReSTOR Aspheric +4 IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- ReSTOR: AcrySof ReSTOR Aspheric +4 Intraocular Lens (IOL)
  Interventions: Device: ReSTOR

INTERVENTIONS:
Device: ReSTOR — Patients were implanted with the AcrySof ReSTOR Aspheric +4 Intraocular Lens (IOL) in one or both eyes for treatment of cataract.

SUMMARY:
To collect visual outcome data post AcrySof ReSTOR Aspheric +4 implantation from surgeons throughout the United States.

ELIGIBILITY:
Inclusion Criteria:

* operable cataracts; candidate for presbyopic correcting intraocular lens (IOL)

Exclusion Criteria:

* ocular comorbidities confounding study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were selected from primary care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2007-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects 18 years of age and older of either sex and any race. Diagnosis of cataracts in one or both eyes.
Pre-assignment Details: Subjects eligibility was determined at the preoperative visit.
Groups:
- ReSTOR: Implantation with the AcrySof ReSTOR Aspheric +4 Intraocular Lens (IOL)
Period: Overall Study
Arm/Group | ReSTOR
Started | 146
Completed | 146
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ReSTOR
Number analyzed (Participants) | 146
Age, Customized [Number; unit: participants] — Age data received on only 124 subjects.
  participants
    <=18 years | 0
    Between 18 and 65 years | 65
    >=65 years | 59
Sex/Gender, Customized [Number; unit: participants] — Gender data received on only 133 subjects
  participants
    Female | 79
    Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Uncorrected Visual Acuity (UCVA) and Best Spectacle Corrected Visual Acuity (BSCVA) at distance (4 meters) and near at preferred distance and measured by logMAR. LogMAR is the "logarithm of the minimum angle of resolution". It is a unit of measure for visual acuity (VA). A lower logMAR value indicates better visual acuity.
Time Frame: 1 week to 10 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR
Number analyzed (Participants) | 146
logMAR
  Distance (4 meters) UCVA | 0.07 (0.12)
  Near (preferred distance) UCVA | 0.07 (0.11)
  Distance (4 meters) BSCVA | 0.02 (0.10)
  Near (preferred distance) BSCVA | 0.06 (0.11)

2. Secondary Outcome: Contrast Sensitivity
Description: Contrast sensitivity is the measurement of how faded an image may become before it is indistinguishable. Contrast sensitivity was measured in photopic, mesopic, and mesopic with glare conditions at the following spatial frequencies: 1.5, 3, 6, 12, and 18 cpd (cycles per degree). Contrast sensitivity is measured in log units. A higher value for the logarithmic units translates to better contrast sensitivity.
Time Frame: 1 week to 10 months
Population: contrast sensitivity data was received for only 51 of 146 patients.
Measure: Mean (Standard Deviation); unit: log units
Arm/Group | ReSTOR
Number analyzed (Participants) | 51
log units
  Photopic condition at 1.5 cpd | 1.61 (0.31)
  Photopic condition at 3 cpd | 1.78 (0.32)
  Photopic condition at 6 cpd | 1.72 (0.44)
  Photopic condition at 12 cpd | 1.22 (0.53)
  Photopic condition at 18 cpd | 0.70 (0.57)
  Mesopic condition at 1.5 cpd | 1.69 (0.30)
  Mesopic condition at 3 cpd | 1.69 (0.32)
  Mesopic condition at 6 cpd | 1.43 (0.57)
  Mesopic condition at 12 cpd | 0.66 (0.67)
  Mesopic condition at 18 cpd | 0.25 (0.45)
  Mesopic with glare condition at 1.5 cpd | 1.29 (0.52)
  Mesopic with glare condition at 3 cpd | 1.28 (0.58)
  Mesopic with glare condition at 6 cpd | 0.92 (0.74)
  Mesopic with glare condition at 12 cpd | 0.27 (0.57)
  Mesopic with glare condition at 18 cpd | 0.07 (0.27)

ADVERSE EVENTS:
Description: Adverse events were not collected for this study because there was no intervention. This was a data collection only study.
Arm/Group | ReSTOR
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor Confidential information will be submitted for publication without Sponsor's prior written agreement.